CLINICAL TRIAL: NCT04245566
Title: Prostatic Artery Embolization vs. Pharmacotherapy for Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia: a Multicenter Randomized Controlled Trial
Brief Title: Prostatic Artery Embolization vs. Pharmacotherapy for LUTS/BPH
Acronym: EMPATHY
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dominik Abt (Other)
Responsible Party: Sponsor-Investigator, Dominik Abt, Principal Investigator, Consultant urologist, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTU19/025
Record Dates: First submitted 2020-01-23; First posted 2020-01-29 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Benign Prostatic Hyperplasia; Pharmacotherapy; Prostatic Artery Embolization; Minimally Invasive Treatment
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: 1:1 randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prostatic Artery Embolization (PAE) (Experimental): PAE will be performed as an inpatient or outpatient procedure by interventional radiologists who are familiar with the procedure and according to established techniques. A unilateral femoral sheath is placed in the right common femoral artery under local anaesthesia. The prostatic arterial supply is identified by selective internal iliac arteriography. Prostatic arteries are selectively catheterised and embolised by use of 250-600 μm microspheres . PAE is performed bilaterally if possible and considered successful in the absence of the normal blush of the prostate and stasis of flow in the prostate arteries on angiography after embolisation.
  Interventions: Procedure: Prostatic Artery Embolization (PAE)
- Pharmocotherapy (Placebo Comparator): Pharmacotherapy will be performed using α1-blockers and 5α-reductase inhibitors in accordance with the EAU recommendations. Thus, patients with a prostate size smaller than 40mL will be treated with 0.4 mg tamsulosin once daily, while patients with larger prostates will be treated with 0.4 mg tamsulosin plus 0.5 mg dutasteride once daily during the complete study follow-up.
  Interventions: Drug: Pharmacotherapy

INTERVENTIONS:
Procedure: Prostatic Artery Embolization (PAE) — Prostatic artery embolization will be performed under local anesthesia according to well established and standardized techniques.
  Arms: Prostatic Artery Embolization (PAE)
Drug: Pharmacotherapy — Pharmacotherapy will be performed using α1-blockers and 5α-reductase inhibitors in accordance with the EAU recommendations
  Arms: Pharmocotherapy

SUMMARY:
This study compares safety and efficacy of prostatic artery embolization and pharmacotherapy in the treatment of lower urinary tract symptoms associated wit benign prostatic hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* men ≥45 years of age
* lower urinary tract symptoms assigned to BPH (diagnosis by medical history and physical examination)
* IPSS ≥ 8 points
* QoL ≥ 3 points
* Qmax ≤ 15 ml/s with a minimum voided volume ≥ 125 ml
* informed consent for study participation

Exclusion Criteria:

* renal impairment (GFR < 30ml/min)
* previous prostatic surgery
* 5-alpha reductase inhibitor (5-ARI) use within 6 mo (or dutasteride within 12 mo) prior to entry, or use of an α-blocker or phytotherapy for BPH within 2 weeks prior to entry
* history or evidence of prostate cancer
* absolute indication for surgical treatment of complications related to BPH (i.e. bladder stones, renal impairment due to bladder outlet obstruction)
* history of neurogenic bladder dysfunction
* not able to complete questionnaires due to cognitive or thought disorders
* language skills insufficient for informed consent and / or completion of questionnaires

Ages: 45 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — based on presence of a prostate
Enrollment: 425 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptoms Score (IPSS) | 24 months after treatment initiation
  The International Prostate Symptoms Score (IPSS) measures the degree of symptoms associated with benign prostatic hyperplasia (BPH). Range of values 0-35 points. Higher values indicate more severe symptoms.

SECONDARY OUTCOMES:
International Prostate Symptoms Score (IPSS) | 6 weeks after treatment initiation
  The International Prostate Symptoms Score (IPSS) measures the degree of symptoms associated with benign prostatic hyperplasia (BPH). Range of values 0-35 points. Higher values indicate more severe symptoms.
International Prostate Symptoms Score (IPSS) | 6 months after treatment initiation
  The International Prostate Symptoms Score (IPSS) measures the degree of symptoms associated with benign prostatic hyperplasia (BPH). Range of values 0-35 points. Higher values indicate more severe symptoms.
International Prostate Symptoms Score (IPSS) | 1 year after treatment initiation
  The International Prostate Symptoms Score (IPSS) measures the degree of symptoms associated with benign prostatic hyperplasia (BPH). Range of values 0-35 points. Higher values indicate more severe symptoms.
International Prostate Symptoms Score (IPSS) | 5 year after treatment initiation
  The International Prostate Symptoms Score (IPSS) measures the degree of symptoms associated with benign prostatic hyperplasia (BPH). Range of values 0-35 points. Higher values indicate more severe symptoms.
Self-assessed goal achievement (SAGA) | 6 weeks after treatment initiation
  SAGA is a PROM focusing on individual treatment goals SAGA is a patient reported outcome measure focusing on individual treatment goals
Self-assessed goal achievement (SAGA) | 6 months after treatment initiation
  SAGA is a PROM focusing on individual treatment goals SAGA is a patient reported outcome measure focusing on individual treatment SAGA is a PROM focusing on individual treatment goals
Self-assessed goal achievement (SAGA) | 1 year after treatment initiation
  SAGA is a PROM focusing on individual treatment goals SAGA is a patient reported outcome measure focusing on individual treatment goals
Self-assessed goal achievement (SAGA) | 2 years after treatment initiation
  SAGA is a PROM focusing on individual treatment goals SAGA is a patient reported outcome measure focusing on individual treatment goals
Self-assessed goal achievement (SAGA) | 5 years after treatment initiation
  SAGA is a PROM focusing on individual treatment goals SAGA is a patient reported outcome measure focusing on individual treatment goals
Maximum urinary stream (Qmax) | 6 weeks after treatment initiation
  Urinary stream will be measured by free uroflowmetry and recorded in mL per second. Higher values indicate a better maximum urinary stream.
Maximum urinary stream (Qmax) | 6 months after treatment initiation
  Urinary stream will be measured by free uroflowmetry and recorded in mL per second. Higher values indicate a better maximum urinary stream.
Maximum urinary stream (Qmax) | 1 year after treatment initiation
  Urinary stream will be measured by free uroflowmetry and recorded in mL per second. Higher values indicate a better maximum urinary stream.
Maximum urinary stream (Qmax) | 2 years after treatment initiation
  Urinary stream will be measured by free uroflowmetry and recorded in mL per second. Higher values indicate a better maximum urinary stream.
Maximum urinary stream (Qmax) | 5 years after treatment initiation
  Urinary stream will be measured by free uroflowmetry and recorded in mL per second. Higher values indicate a better maximum urinary stream.
Post void residual urine (PVR) | 6 weeks after treatment initiation
  Post void residual is measured after voiding by transabdominal ultrasound and calculated in mL. Higher values indicate more post void residual urine and a worse ability to empty the bladder.
Post void residual urine (PVR) | 6 months after treatment initiation
  Post void residual is measured after voiding by transabdominal ultrasound and calculated in mL. Higher values indicate more post void residual urine and a worse ability to empty the bladder.
Post void residual urine (PVR) | 1 year after treatment initiation
  Post void residual is measured after voiding by transabdominal ultrasound and calculated in mL. Higher values indicate more post void residual urine and a worse ability to empty the bladder.
Post void residual urine (PVR) | 2 years after treatment initiation
  Post void residual is measured after voiding by transabdominal ultrasound and calculated in mL. Higher values indicate more post void residual urine and a worse ability to empty the bladder.
Post void residual urine (PVR) | 5 years after treatment initiation
  Post void residual is measured after voiding by transabdominal ultrasound and calculated in mL. Higher values indicate more post void residual urine and a worse ability to empty the bladder.
Prostate volume | 6 moths after treatment initiation
  Prostate volume measured by transrectal ultrasound. This examination is only performed at selected food-up visits (i.e. 6mo, 2y, 5y)
Prostate volume | 2 years after treatment initiation
  Prostate volume measured by transrectal ultrasound. This examination is only performed at selected food-up visits (i.e. 6mo, 2y, 5y)
Prostate volume | 5 years after treatment initiation
  Prostate volume measured by transrectal ultrasound. This examination is only performed at selected food-up visits (i.e. 6mo, 2y, 5y)
Prostate specific antigen (PSA) | 6 months after treatment initiation
  laboratory test
Prostate specific antigen (PSA) | 1 year after treatment initiation
  laboratory test
Prostate specific antigen (PSA) | 2 years after treatment initiation
  laboratory test
Prostate specific antigen (PSA) | 5 years after treatment initiation
  laboratory test
Safety / adverse events | 6 weeks after treatment initiation
  Number of patients developing adverse events: Classification will be performed according to Clavien-Dindo classification and CTCAE.
Safety / adverse events | 6 months after treatment initiation
  Number of patients developing adverse events: Classification will be performed according to Clavien-Dindo classification and CTCAE.
Safety / adverse events | 1 year after treatment initiation
  Number of patients developing adverse events: Classification will be performed according to Clavien-Dindo classification and CTCAE.
Safety / adverse events | 2 year after treatment initiation
  Number of patients developing adverse events: Classification will be performed according to Clavien-Dindo classification and CTCAE.
Safety / adverse events | 5 year after treatment initiation
  Number of patients developing adverse events: Classification will be performed according to Clavien-Dindo classification and CTCAE.
Erectile function | 6 weeks after treatment initiation
  Assessed by the questionnaire IIEF-5. Score of IIEF-5 can range from 0 to 25 points. Higher values indicate a better erectile function.
Erectile function | 6 months after treatment initiation
  Assessed by the questionnaire IIEF-5. Score of IIEF-5 can range from 0 to 25 points. Higher values indicate a better erectile function.
Erectile function | 1 year after treatment initiation
  Assessed by the questionnaire IIEF-5. Score of IIEF-5 can range from 0 to 25 points. Higher values indicate a better erectile function.
Erectile function | 2 year after treatment initiation
  Assessed by the questionnaire IIEF-5. Score of IIEF-5 can range from 0 to 25 points. Higher values indicate a better erectile function.
Erectile function | 5 year after treatment initiation
  Assessed by the questionnaire IIEF-5. Score of IIEF-5 can range from 0 to 25 points. Higher values indicate a better erectile function.
Ejaculatory function | 6 weeks after treatment initiation
  Assessed by the questionnaire Male Sexual Health Questionnaire-Ejaculation Dysfunction Short Form (MSHQ-EjD). Ejaculatory function total score (questions 1-3, possible range 0-15, higher values indicate better ejaculatory function, and MSHQ-EjD ejaculatory bother item (question 4, possible range 0-5, higher values indicate more bother).
Ejaculatory function | 6 months after treatment initiation
  Assessed by the questionnaire Male Sexual Health Questionnaire-Ejaculation Dysfunction Short Form (MSHQ-EjD). Ejaculatory function total score (questions 1-3, possible range 0-15, higher values indicate better ejaculatory function, and MSHQ-EjD ejaculatory bother item (question 4, possible range 0-5, higher values indicate more bother).
Ejaculatory function | 1 year after treatment initiation
  Assessed by the questionnaire Male Sexual Health Questionnaire-Ejaculation Dysfunction Short Form (MSHQ-EjD). Ejaculatory function total score (questions 1-3, possible range 0-15, higher values indicate better ejaculatory function, and MSHQ-EjD ejaculatory bother item (question 4, possible range 0-5, higher values indicate more bother).
Ejaculatory function | 2 years after treatment initiation
  Assessed by the questionnaire Male Sexual Health Questionnaire-Ejaculation Dysfunction Short Form (MSHQ-EjD). Ejaculatory function total score (questions 1-3, possible range 0-15, higher values indicate better ejaculatory function, and MSHQ-EjD ejaculatory bother item (question 4, possible range 0-5, higher values indicate more bother).
Ejaculatory function | 5 years after treatment initiation
  Assessed by the questionnaire Male Sexual Health Questionnaire-Ejaculation Dysfunction Short Form (MSHQ-EjD). Ejaculatory function total score (questions 1-3, possible range 0-15, higher values indicate better ejaculatory function, and MSHQ-EjD ejaculatory bother item (question 4, possible range 0-5, higher values indicate more bother).
Need for additional drug treatment, surgical treatment or change of medical treatment assessed | 6 weeks after treatment initiation
  assessed by patient interviews at follow up visit
Need for additional drug treatment, surgical treatment or change of medical treatment assessed | 6 moths after treatment initiation
  assessed by patient interviews at follow up visit
Need for additional drug treatment, surgical treatment or change of medical treatment assessed | 1 year after treatment initiation
  assessed by patient interviews at follow up visit
Need for additional drug treatment, surgical treatment or change of medical treatment assessed | 2 years after treatment initiation
  assessed by patient interviews at follow up visit
Need for additional drug treatment, surgical treatment or change of medical treatment assessed | 5 years after treatment initiation
  assessed by patient interviews at follow up visit
Analysis of cost-effectiveness using quality-adjusted life years (QALY) | 2 years after treatment initiation
  One QALY equates to one year in perfect health. QALY scores range from 1 (perfect health) to 0 (dead). To estimate QALY costs will be calculated by calculation of treatment costs, and quality of life will be assessed using the questionnaire EQ-5D. EQ-5D measures five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Respondents self-rate their level of severity for each dimension using a five-level scale. The questionnaire can define 3,125 different health states.
Analysis of cost-effectiveness using quality-adjusted life years (QALY) | 5 years after treatment initiation
  One QALY equates to one year in perfect health. QALY scores range from 1 (perfect health) to 0 (dead). To estimate QALY costs will be calculated by calculation of treatment costs, and quality of life will be assessed using the questionnaire EQ-5D. EQ-5D measures five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Respondents self-rate their level of severity for each dimension using a five-level scale. The questionnaire can define 3,125 different health states.

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Abt, MD, Principal Investigator — Cantonal Hospital of St. Gallen

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, data are stored in a publicly accessible repository (e.g.
  Harvard Dataverse or Zenodo, depending on whether the data should be stored on a server in America or Europe). All elements are stored with a unique Digital Object Identifier (DOI), which can be referenced in the respective publication.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: At the end of the study. Availability for at least 10 years.